CLINICAL TRIAL: NCT00207714
Title: A Randomized, Double-blind, Dose-ranging Trial of CNTO 148 Subcutaneous Injection Compared With Placebo in Subjects With Active Rheumatoid Arthritis Despite Treatment With Methotrexate
Brief Title: An Efficacy and Safety Study of CNTO 148 Subcutaneous Injection Compared With Placebo in Patients With Active Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centocor, Inc. (Industry)
Collaborators: Centocor BV (Industry)
Responsible Party: DIRECTOR CLINICAL RESEARCH, Janssen R&D US
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR005263; C0524T02 (Other: Centocor)
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Results first posted 2012-08-07 (Estimated); Last update posted 2012-10-18 (Estimated); Status verified 2012-10

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; CNTO 148; Methotrexate; Joint pain; Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthralgia; Arthritis | interventions — golimumab; Infliximab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Golimumab (CNTO 148) with Methotrexate (MTX) (Experimental)
  Interventions: Drug: Golimumab; Drug: MTX
- Infliximab with MTX (Experimental)
  Interventions: Drug: MTX; Drug: Infliximab
- Placebo with MTX (Placebo Comparator)
  Interventions: Drug: MTX; Drug: Placebo

INTERVENTIONS:
Drug: Golimumab — Type=exact, unit=mg/ml, number= 50 to 100 , form=powder for solution for infusion, route=sub cutaneous.
  Arms: Golimumab (CNTO 148) with Methotrexate (MTX)
Drug: MTX — Type=exact, unit=mg/ml, number= 10, form=powder for solution for infusion, route=sub cutaneous
Drug: Placebo — Type=exact, unit=mg/ml, form=powder for solution for infusion, route=sub cutaneous
  Arms: Placebo with MTX
Drug: Infliximab — Type=exact, unit=mg/ml number= 10, form=powder for solution for infusion, route=sub cutaneous
  Arms: Infliximab with MTX

SUMMARY:
Multicenter, randomized, double-blind, placebo-controlled, 5-arm, dose-ranging study to assess the efficacy of subcutaneous injections of Golimumab (CNTO 148), 50 or 100 mg, at either 2- or 4- week intervals in subjects with active RA despite MTX therapy.

DETAILED DESCRIPTION:
This is an experimental medical research study. The purpose of this study is to determine if Golimumab is safe and effective in the treatment of rheumatoid arthritis.

Subjects will receive subcutaneous injections of either 50 or 100 mg Golimumab or placebo every two or four weeks or an infusion of infliximab at week 20, 22, 28, 36, 44 for 48 weeks

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of RA according to the American College of Rheumatology criteria for at least 3 months prior to screening
* Have active Rheumatoid Arthritis at the time of screening and at baseline, as defined by 6 or more swollen joints and 6 or more tender joints and additional laboratory criteria

Exclusion Criteria:

* Have other inflammatory diseases, including but not limited to ankylosing spondylitis, systemic lupus erythematosus, Lyme disease
* Received disease-modifying antirheumatic drugs ([DMARDs] eg, D penicillamine, hydroxychloroquine, chloroquine, oral or parenteral gold, interleukin [IL]-1 receptor antagonist [anakinra], azathioprine, sulphasalazine, agents other than MTX) within 4 weeks prior to the first study dose

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2003-11; Primary Completion 2005-02 (Actual); Study Completion 2006-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.

REFERENCES:
- [Derived] Kay J, Matteson EL, Dasgupta B, Nash P, Durez P, Hall S, Hsia EC, Han J, Wagner C, Xu Z, Visvanathan S, Rahman MU. Golimumab in patients with active rheumatoid arthritis despite treatment with methotrexate: a randomized, double-blind, placebo-controlled, dose-ranging study. Arthritis Rheum. 2008 Apr;58(4):964-75. doi: 10.1002/art.23383. PMID 18383539

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 172 participants were randomly assigned to treatments at 33 sites: 16 in North America (13 in the US and 3 in Canada), 12 in Europe (3 in Belgium, 4 in the UK, 5 in Germany), and 5 in Australia. The study period extended from 01 Dec 2003 to 21 Feb 2006.
Groups:
- Group I: Placebo Crossover to Infliximab: Placebo subcutaneous (SC) injections every 2 weeks (Wks) from Week (Wk) 0 thru Wk 18 plus Methotrexate (MTX) (Wks 0, 2, 4, 6, 8, 10, 12, 14, 16, and 18); after all study evaluations at Wk 20, open-label infliximab intravenous (IV) infusions: 3 milligrams per kilogram (mg/kg) at Wks 20, 22, 28 and then every 8 Wks thru Wk 44. Continue stable dose of MTX throughout the study.
- Group II: Golimumab 50 mg Every 4 Weeks: Golimumab (CNTO148) 50 milligram (mg) SC injections every 4 Wks from Wk 0 thru Wk 18 plus MTX (Wks 0, 4, 8, 12, and 16); Placebo SC injections were to be administered at interim visits (Wks 2, 6, 10, 14, and 18) plus MTX. Participants continued at 50 mg of golimumab at Wk 20, and then every 4 Wks thru Wk 48. Continue stable dose of MTX throughout the study. Participants remained blinded thru the end of study. Also referred to as Group II: golimumab 50 mg plus placebo every 4 Wks.
- Group III: Golimumab 50 mg Every 2 or 4 Weeks: Golimumab 50 mg SC injections every 2 Wks from Wk 0 thru Wk 18 plus MTX (Wks 0, 2, 4, 6, 8, 10, 12, 14, 16, and 18); Participants continued at 50 mg of golimumab at Wk 20, and then every 4 Wks through Wk 48. Continue stable dose of MTX throughout the study. Participants remained blinded thru the end of study. Also referred to as GroupIII: Golimumab 50 mg every 2 or 4 Wks.
- Group IV: Golibumab 100 mg Every 4 Weeks: Golimumab 100 mg SC injections every 4 Wks thru Wk 18 plus MTX (Wks 0, 4, 8, 12, and 16); Placebo SC injections were to be administered at interim visits (Wks 2, 6, 10, 14, and 18) plus MTX. Participants continued at 100 mg of golimumab at Wk 20, and then every 4 Wks through Wk 48. Continue stable dose of MTX throughout the study. Participants remained blinded through the end of study. Also referred to as Group IV: golimumab 100 mg plus placebo every 4 Wks.
- Group V: Golimumab 100 mg Every 2 or 4 Weeks: Golimumab 100 mg SC injections every 2 Wks from Wk 0 thru Wk 18 plus MTX (Wks 0, 2, 4, 6, 8, 10, 12, 14, 16, and 18); Participants continued at 100 mg of golimumab at Wk 20, and then every 4 Wks through Wk 48. Continue stable dose of MTX throughout the study. Participants remained blinded thru the end of study. Also referred to as Group V: Golimumab 100 mg every 2 or 4 Wks.
Period: Overall Study
Arm/Group | Group I: Placebo Crossover to Infliximab | Group II: Golimumab 50 mg Every 4 Weeks | Group III: Golimumab 50 mg Every 2 or 4 Weeks | Group IV: Golibumab 100 mg Every 4 Weeks | Group V: Golimumab 100 mg Every 2 or 4 Weeks
Started | 35 | 35 | 34 | 34 | 34
Completed | 21 (Indicates number of participants who continued subcutaneous study agent at Wk 16) | 28 (Indicates number of participants who continued subcutaneous study agent at Wk 16) | 24 (Indicates number of participants who continued subcutaneous study agent at Wk 16) | 26 (Indicates number of participants who continued subcutaneous study agent at Wk 16) | 29 (Indicates number of participants who continued subcutaneous study agent at Wk 16)
Not Completed | 14 | 7 | 10 | 8 | 5
Not completed — Adverse Event | 6 | 2 | 4 | 3 | 1
Not completed — Unsatisfactory therapeutic effect | 5 | 3 | 1 | 4 | 4
Not completed — Other | 3 | 2 | 5 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group I: Placebo Crossover to Infliximab | Group II: Golimumab 50 mg Every 4 Weeks | Group III: Golimumab 50 mg Every 2 or 4 Weeks | Group IV: Golibumab 100 mg Every 4 Weeks | Group V: Golimumab 100 mg Every 2 or 4 Weeks | Total
Number analyzed (Participants) | 35 | 35 | 34 | 34 | 34 | 172
Age Continuous [Mean (Standard Deviation); unit: Years] | 53.8 (12.9) | 56.1 (10.5) | 50.4 (13.1) | 56.3 (12.1) | 54.1 (14.1) | 54.2 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 30 | 23 | 26 | 27 | 132
  Male | 9 | 5 | 11 | 8 | 7 | 40

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Meeting the American College of Rheumatology 20 (ACR 20) Response at Week 16
Description: ACR 20 response is a decrease of at least 20 per cent in both tender and swollen joint count and in 3 to 5 assessments (participant's assessment of pain visual analog scale [VAS] with 0, no pain to 10, worst pain; patient's and physician's global assessment of disease activity VAS scales: overall disease activity [0, very well to 10, very poor and 0, no arthritis activity to 10, extremely active, respectively]; Health Assessment Questionnaire [HAQ]: 20-questions on life activities [0, no difficulty to 3, inability to perform a task]; C-reactive protein[CRP]).
Time Frame: Week 16
Population: Intent to treat (ITT). Participants considered non-responder if used any pre-specified prohibited medications or discontinued subcutaneous (SC) study agent due to lack of efficacy. Missing ACR components were imputed by Last Observation Carried Forward (LOCF) unless all ACR components are missing in which case considered non-responders.
Measure: Number; unit: Participants
Groups:
- Group I: Placebo Crossover to Infliximab: Placebo SC injections every 2 weeks (Wks) from week (Wk) 0 thru Wk 18 plus Methotrexate (MTX) (Wks 0, 2, 4, 6, 8, 10, 12, 14, 16, and 18); after all study evaluations at Wk 20, open-label infliximab IV infusions: 3 mg/kg at Wks 20, 22, 28 and then every 8 Wks thru Wk 44. Continue stable dose of MTX throughout the study.
- Group II: Golimumab 50 mg Every 4 Weeks: Golimumab (CNTO148) 50 mg SC injections every 4 Wks from Wk 0 thru Wk 18 plus MTX (Wks 0, 4, 8, 12, and 16); Placebo SC injections were to be administered at interim visits (Wks 2, 6, 10, 14, and 18) plus MTX. Participants continued at 50 mg of golimumab at Wk 20, and then every 4 Wks thru Wk 48. Continue stable dose of MTX throughout the study. Participants remained blinded thru the end of study.
- Group III: Golimumab 50 mg Every 2 or 4 Weeks: Golimumab 50 mg SC injections every 2 Wks from Wk 0 thru Wk 18 plus MTX (Wks 0, 2, 4, 6, 8, 10, 12, 14, 16, and 18); Participants continued at 50 mg of golimumab at Wk 20, and then every 4 Wks through Wk 48. Continue stable dose of MTX throughout the study. Participants remained blinded thru the end of study.
- Group IV: Golibumab 100 mg Every 4 Weeks: Golimumab 100 mg SC injections every 4 Wks thru Wk 18 plus MTX (Wks 0, 4, 8, 12, and 16); Placebo SC injections were to be administered at interim visits (Wks 2, 6, 10, 14, and 18) plus MTX. Participants continued at 100 mg of golimumab at Wk 20, and then every 4 Wks through Wk 48. Continue stable dose of MTX throughout the study. Participants remained blinded through the end of study.
- Group V: Golimumab 100 mg Every 2 or 4 Weeks: Golimumab 100 mg SC injections every 2 Wks from Wk 0 thru Wk 18 plus MTX (Wks 0, 2, 4, 6, 8, 10, 12, 14, 16, and 18); Participants continued at 100 mg of golimumab at Wk 20, and then every 4 Wks through Wk 48. Continue stable dose of MTX throughout the study. Participants remained blinded thru the end of study.
- Combined: Groups II, III, IV & V: Combines Groups II (golimumab 50 mg plus placebo), III (golimumab 50 mg every 2/4 Wks), IV (golimumab 100 mg plus placebo) & V (golimumab 100 mg every 2/4 Wks).
Arm/Group | Group I: Placebo Crossover to Infliximab | Group II: Golimumab 50 mg Every 4 Weeks | Group III: Golimumab 50 mg Every 2 or 4 Weeks | Group IV: Golibumab 100 mg Every 4 Weeks | Group V: Golimumab 100 mg Every 2 or 4 Weeks | Combined: Groups II, III, IV & V
Number analyzed (Participants) | 35 | 35 | 34 | 34 | 34 | 137
Participants | 13 | 21 | 17 | 19 | 27 | 84
Statistical Analysis 1: Comparison: Group I: Placebo Crossover to Infliximab vs Combined: Groups II, III, IV & V; Null hypothesis: No difference in ACR 20 response at Week 16 between combined golimumab groups and Placebo +MTX group. Sample of 35 participants per treatment groups (140 in combined golimumab group and 35 in Placebo +MTX group) provides greater than 90% power assuming 60% golimumab response and 25 % response in Placebo +MTX; Test type: Superiority or Other; p = 0.010, Cochran-Mantel-Haenszel — A positive test is concluded if there is a significant difference between combined golimumab and placebo groups and at least one of the pair-wise comparisons at 0.05 level
Statistical Analysis 2: Comparison: Group I: Placebo Crossover to Infliximab vs Group II: Golimumab 50 mg Every 4 Weeks; Null hypothesis: No difference in ACR 20 response at Wk 16 between golimumab 50 mg every 4 weeks and Placebo + MTX. Sample of 35 participants per treatment groups (140 in combined golimumab group and 35 in Placebo +MTX group) provides greater than 90% power assuming 60% golimumab response and 25% response in placebo; Test type: Superiority or Other; p = 0.056, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Group I: Placebo Crossover to Infliximab vs Group III: Golimumab 50 mg Every 2 or 4 Weeks; Null hypothesis: No difference in ACR 20 response at Wk 16 between Golimumab 50 mg every 2 or 4 Weeks and Placebo + MTX. Sample of 35 participants per treatment groups (140 in combined golimumab group and 35 in Placebo +MTX group) provides greater than 90% power assuming 60% golimumab response and 25% response in placebo; Test type: Superiority or Other; p = 0.281, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Group I: Placebo Crossover to Infliximab vs Group IV: Golibumab 100 mg Every 4 Weeks; Null hypothesis: No difference in ACR 20 response at Wk 16 between Golimumab 100 mg every 4 weeks and Placebo + MTX. Sample of 35 participants per treatment groups (140 in combined golimumab group and 35 in Placebo +MTX group) provides greater than 90% power assuming 60% golimumab response and 25% response in placebo; Test type: Superiority or Other; p = 0.119, Cochran-Mantel-Haenszel
Statistical Analysis 5: Comparison: Group I: Placebo Crossover to Infliximab vs Group V: Golimumab 100 mg Every 2 or 4 Weeks; Null hypothesis: No difference in ACR 20 response at Wk 16 between Golimumab 100 mg every 2 or 4 Weeks and Placebo + MTX. Sample of 35 participants per treatment groups (140 in combined golimumab group and 35 in Placebo +MTX group) provides greater than 90% power assuming 60% golimumab response and 25% response in placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

2. Secondary Outcome: Summary of ACR-N, Index of Improvement at Week 16
Description: The ACR-N index of improvement is the minimum of the following: 1) the percent decrease from baseline in tender joint counts; 2) the percent decrease from baseline in swollen joint counts; 3) the median percent decrease from baseline for the following: a. Patient's assessment of pain as measured on a 10 cm visual assessment scale (0-10, 10 worst pain) Patient's global assessment of disease activity (VAS 0-10); c. Physician's global assessment of disease activity (VAS 0-10) d. Physical function as measured by the Health Assessment Questionnaire; e. C-Reactive Protein measurement.
Time Frame: Week 16
Population: Intent-to-treat (ITT) and missing ACR components were imputed by LOCF unless all ACR components are missing in which case considered non-responders. The joint evaluability rules were also applied.
Measure: Median (Inter-Quartile Range); unit: Scores on scale
Groups:
- Group I: Placebo Crossover to Infliximab: Placebo SC injections every 2 wks from Wk 0 thru Wk 18 plus Methotrexate (MTX) (Wks 0, 2, 4, 6, 8, 10, 12, 14, 16, and 18); after all study evaluations at Wk 20, open-label infliximab IV infusions: 3 mg/kg at Wks 20, 22, 28 and then every 8 wks thru Wk 44. Continue stable dose of MTX throughout the study.
- Group III: Golimumab 50 mg Every 2 or 4 Weeks: Golimumab 50 mg SC injections every 2 wks from Wk 0 thru Wk 18 plus MTX (Wks 0, 2, 4, 6, 8, 10, 12, 14, 16, and 18); Participants continued at 50 mg of golimumab at Wk 20, and then every 4 weeks through Wk 48. Continue stable dose of MTX throughout the study. Participants remained blinded thru the end of study.
- Group IV: Golibumab 100 mg Every 4 Weeks: Golimumab 100 mg SC injections every 4 wks thru Wk 18 plus MTX (Weeks 0, 4, 8, 12, and 16); Placebo SC injections were to be administered at interim visits (Weeks 2, 6, 10, 14, and 18) plus MTX. Participants continued at 100 mg of golimumab at Wk 20, and then every 4 wks through Wk 48. Continue stable dose of MTX throughout the study. Participants remained blinded through the end of study.
- Group V: Golimumab 100 mg Every 2 or 4 Weeks: Golimumab 100 mg SC injections every 2 wks from Wk 0 thru Wk 18 plus MTX (Wks 0, 2, 4, 6, 8, 10, 12, 14, 16, and 18); Participants continued at 100 mg of golimumab at Wk 20, and then every 4 weeks through Wk 48. Continue stable dose of MTX throughout the study. Participants remained blinded thru the end of study.
Arm/Group | Group I: Placebo Crossover to Infliximab | Group II: Golimumab 50 mg Every 4 Weeks | Group III: Golimumab 50 mg Every 2 or 4 Weeks | Group IV: Golibumab 100 mg Every 4 Weeks | Group V: Golimumab 100 mg Every 2 or 4 Weeks | Combined: Groups II, III, IV & V
Number analyzed (Participants) | 35 | 35 | 34 | 34 | 34 | 137
Scores on scale | 0.0 [-12.5 to 28.6] | 37.4 [0.0 to 54.4] | 19.4 [-1.0 to 49.0] | 22.3 [0.0 to 55.6] | 35.6 [20.0 to 56.6] | 33.3 [0.0 to 54.4]
Statistical Analysis 1: Comparison: Group I: Placebo Crossover to Infliximab vs Combined: Groups II, III, IV & V; No difference in ACRn scores measured as percentage of improvement from baseline at Week 16 between Placebo + MTX and combined golimumab groups; Test type: Superiority or Other; p = 0.001, ANOVA on van der Waerden normal scores
Statistical Analysis 2: Comparison: Group I: Placebo Crossover to Infliximab vs Group II: Golimumab 50 mg Every 4 Weeks; No difference in ACRn scores measured as percentage of improvement from baseline at Week 16 between Placebo + MTX and Golimumab 50 mg every 4 weeks; Test type: Superiority or Other; p = 0.006, ANOVA on van der Waerden normal scores
Statistical Analysis 3: Comparison: Group I: Placebo Crossover to Infliximab vs Group III: Golimumab 50 mg Every 2 or 4 Weeks; No difference in ACRn scores measured as percentage of improvement from baseline at Week 16 between Placebo + MTX and Golimumab 50 mg every 2 or 4 Weeks; Test type: Superiority or Other; p = 0.095, ANOVA on van der Waerden normal scores
Statistical Analysis 4: Comparison: Group I: Placebo Crossover to Infliximab vs Group IV: Golibumab 100 mg Every 4 Weeks; No difference in ACRn scores measured as percentage of improvement from baseline at Week 16 between Placebo + MTX Golibumab 100 mg every 4 weeks; Test type: Superiority or Other; p = 0.010, ANOVA on van der Waerden normal scores; ANOVA on van der Waerden normal scores
Statistical Analysis 5: Comparison: Group I: Placebo Crossover to Infliximab vs Group V: Golimumab 100 mg Every 2 or 4 Weeks; No difference in ACRn scores measured as percentage of improvement from baseline at Week 16 between Placebo + MTX Golimumab 100 mg every 2 or 4 Weeks; Test type: Superiority or Other; p < 0.001, ANOVA on van der Waerden normal scores

ADVERSE EVENTS:
Time Frame: Baseline to Week 52
Description: Twelve participants received an incorrect study agent or incorrect dose of Golimumab (CNTO 148) at least once through Week 16. For analyses performed by actual treatment received, 10 subjects were counted in treatment groups (based on total dose received) that differed from the treatment groups to which they had been randomly assigned.
Groups:
- Group II: Golimumab 50 mg Every 4 Weeks: Golimumab (CNTO148) 50 milligram (mg) subcutaneous (SC) injections every 4 weeks (Wks) from Week (Wk) 0 thru Wk 18 plus methotrexate (MTX) (Wks 0, 4, 8, 12, and 16); Placebo SC injections were to be administered at interim visits (Wks 2, 6, 10, 14, and 18) plus MTX. Patients continued at 50 mg of golimumab at Wk 20, and then every 4 Wks thru Wk 48. Continue stable dose of MTX throughout the study. Patients remained blinded thru the end of study. Also referred to as Group II: golimumab 50 mg plus placebo every 4 Wks.
- Group III: Golimumab 50 mg Every 2 or 4 Weeks: Golimumab 50 miligram (mg) subcutaneous (SC) injections every 2 weeks (Wks) from Week (Wk) 0 thru Wk 18 plus methotrexate (MTX) (Wks 0, 2, 4, 6, 8, 10, 12, 14, 16, and 18); Patients continued at 50 mg of golimumab at Wk 20, and then every 4 Wks through Wk 48. Continue stable dose of MTX throughout the study. Patients remained blinded thru the end of study. Also referred to as GroupIII: Golimumab 50 mg every 2 or 4 Wks.
- Group IV: Golibumab 100 mg Every 4 Weeks: Golimumab 100 mg subcutaneous (SC) injections every 4 weeks (Wks) thru Week (Wk) 18 plus methotrexate (MTX) (Wks 0, 4, 8, 12, and 16); Placebo SC injections were to be administered at interim visits (Wks 2, 6, 10, 14, and 18) plus MTX. Patients continued at 100 mg of golimumab at Wk 20, and then every 4 Wks through Wk 48. Continue stable dose of MTX throughout the study. Patients remained blinded through the end of study. Also referred to as Group IV: golimumab 100 mg plus placebo every 4 Wks.
- Group V: Golimumab 100 mg Every 2 or 4 Weeks: Golimumab 100 milligrams (mg) subcutaneous (SC) injections every 2 weeks (Wks) from Week (Wk) 0 thru Wk 18 plus methotrexate (MTX) (Wks 0, 2, 4, 6, 8, 10, 12, 14, 16, and 18); Patients continued at 100 mg of golimumab at Wk 20, and then every 4 Wks through Wk 48. Continue stable dose of MTX throughout the study. Patients remained blinded thru the end of study. Also referred to as Group V: Golimumab 100 mg every 2 or 4 Wks.
Arm/Group | Group I: Placebo Crossover to Infliximab | Group II: Golimumab 50 mg Every 4 Weeks | Group III: Golimumab 50 mg Every 2 or 4 Weeks | Group IV: Golibumab 100 mg Every 4 Weeks | Group V: Golimumab 100 mg Every 2 or 4 Weeks
Serious Adverse Events (participants affected / at risk) | 2/34 | 7/37 | 5/32 | 5/33 | 5/35
Other Adverse Events (participants affected / at risk) | 28/34 | 34/37 | 29/32 | 29/33 | 33/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group I: Placebo Crossover to Infliximab (N=34) | Group II: Golimumab 50 mg Every 4 Weeks (N=37) | Group III: Golimumab 50 mg Every 2 or 4 Weeks (N=32) | Group IV: Golibumab 100 mg Every 4 Weeks (N=33) | Group V: Golimumab 100 mg Every 2 or 4 Weeks (N=35)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Fracture delayed union (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Bronchopneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pneumonia legionella (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Listeria sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Fractured coccyx (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Medical device complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Chronic obstructive airways disease exacerbated (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Thrombophlebitis superficial (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Nerve root compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group I: Placebo Crossover to Infliximab (N=34) | Group II: Golimumab 50 mg Every 4 Weeks (N=37) | Group III: Golimumab 50 mg Every 2 or 4 Weeks (N=32) | Group IV: Golibumab 100 mg Every 4 Weeks (N=33) | Group V: Golimumab 100 mg Every 2 or 4 Weeks (N=35)
Nasopharyngitis (Infections and infestations) | 3 | 8 | 3 | 2 | 8
Upper respiratory tract infection (Infections and infestations) | 7 | 6 | 6 | 5 | 4
Influenza (Infections and infestations) | 0 | 4 | 2 | 2 | 1
Sinusitis (Infections and infestations) | 2 | 3 | 3 | 2 | 1
Bronchitis (Infections and infestations) | 1 | 3 | 0 | 0 | 5
Herpes simplex (Infections and infestations) | 1 | 3 | 2 | 1 | 1
Urinary tract infection (Infections and infestations) | 2 | 2 | 0 | 3 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 1 | 1 | 2 | 1
Lower respiratory tract infection (Infections and infestations) | 3 | 1 | 0 | 3 | 1
Respiratory tract infection (Infections and infestations) | 1 | 3 | 1 | 1 | 0
Viral infection (Infections and infestations) | 0 | 2 | 1 | 1 | 1
Pharyngitis (Infections and infestations) | 0 | 2 | 0 | 1 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 1 | 0 | 3
Nail infection (Infections and infestations) | 0 | 0 | 2 | 1 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0
Fungal rash (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Gingival infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 5 | 8 | 7 | 4 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 5 | 2 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 3 | 2 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 3 | 2 | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3 | 1 | 3
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 0 | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 2
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 0 | 0
Shoulder pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 2
Injection site erythema (General disorders) | 4 | 5 | 5 | 4 | 10
Fatigue (General disorders) | 0 | 2 | 4 | 2 | 3
Pyrexia (General disorders) | 1 | 3 | 1 | 4 | 2
Injection site pain (General disorders) | 0 | 1 | 2 | 3 | 2
Oedema peripheral (General disorders) | 0 | 3 | 3 | 1 | 1
Chest pain (General disorders) | 0 | 0 | 2 | 1 | 3
Injection site pruritus (General disorders) | 0 | 1 | 0 | 1 | 3
Chills (General disorders) | 2 | 0 | 1 | 2 | 1
Injection site induration (General disorders) | 0 | 1 | 1 | 0 | 2
Malaise (General disorders) | 0 | 2 | 0 | 1 | 1
Injection site haemorrhage (General disorders) | 1 | 0 | 2 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 5 | 8 | 7 | 8
Diarrhoea (Gastrointestinal disorders) | 4 | 5 | 3 | 3 | 6
Vomiting (Gastrointestinal disorders) | 2 | 5 | 0 | 2 | 5
Abdominal pain upper (Gastrointestinal disorders) | 4 | 2 | 2 | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 1
Constipation (Gastrointestinal disorders) | 1 | 2 | 1 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 4 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 1
Gingival pain (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Headache (Nervous system disorders) | 7 | 8 | 6 | 9 | 3
Dizziness (Nervous system disorders) | 6 | 1 | 3 | 4 | 3
Paraesthesia (Nervous system disorders) | 0 | 3 | 2 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 1 | 1 | 2
Sciatica (Nervous system disorders) | 0 | 3 | 0 | 1 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 5 | 4 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 3 | 2
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 3 | 2 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0 | 0
Rhinitis seasonal (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 2 | 0 | 1 | 3
Rash (Skin and subcutaneous tissue disorders) | 3 | 2 | 1 | 1 | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 3 | 1 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 3 | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 0 | 0
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 2 | 2
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 1 | 2
Excoriation (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 2 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 4 | 3 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 3 | 3 | 1
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 1 | 2
Blood pressure increased (Investigations) | 0 | 0 | 0 | 2 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 2 | 0
Hypertension (Vascular disorders) | 1 | 4 | 3 | 1 | 2
Hot flush (Vascular disorders) | 2 | 1 | 2 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 2 | 1 | 2
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 2 | 0
Dry eye (Eye disorders) | 1 | 0 | 0 | 2 | 1
Conjunctivitis (Eye disorders) | 1 | 2 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 2 | 0 | 0
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 0
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
The count of patients with any nonserious adverse events (NAE) excludes patients who only had NAE that occurred in <= 5% of patients. This information may vary from existing approved labeling and publications due to the requirement of this website.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Generally, the only disclosure restriction on the Principal Investigator is that the sponsor has 60 days to review results communications prior to public release and can embargo communications regarding trial results for a period that does not exceed 180 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.